CLINICAL TRIAL: NCT05135416
Title: The Impact of Chewing Gum on Postoperative Bowel Activity and Postoperative Pain After Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ŞENAY DEMİRBAŞ MEYDAN, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 1111
Record Dates: First submitted 2021-09-29; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Postoperative Pain
Keywords: Pain; Total Laparoscopic Hysterectomy Surgery; Bowel Functions; Chewing Gum; Nursing
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: crossover assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chewing gum Group (Active Comparator): Questions related to surgery and bowel function found in the Participant Information Form it will be filled in. The chewing gum group data will be followed up with the "Follow-up Form- Chewing Gum Group ". Women who make up the gum group, based on the time of arrival in the room 2. per hour, 4. and 6 o'clock. they'll chew gum an hour. Chewing gum based on knowledge of the literature its duration will be limited to 15 minutes, and a new gum will be introduced with each chewing. To all women the same brand will be given unsweetened chewing gum, which is easy to chew, does not contain sorbitol and xylitol. Sorbitol GIS problems in the case of ingestion of gums containing it, while gums containing xylitol are more in order not to ignore the decongestant risk of diarrhea when consumed, sugar-free chewing gum was preferred.
  Interventions: Procedure: chewing gum Group
- Control group (Active Comparator): Questions related to surgery and bowel function found in the Participant Information Form it will be filled in. The control group data were followed up with the "Follow-up Form-Control Group" will be. Of the women who made up the control group, it was not until the bowel sounds were first heard that bowel sounds will be listened to by the service nurse december 2 hours intervals. The patient has gas-stool by querying the output, it will be saved. Application of analgesics to pain levelsin the case of "Visual Analog Scale" (Visual Analog Scale -Vas) within 15 minutes it will be evaluated with. After the end of the researcher's 8-hour shift, the time of gas extraction and defecation is estimated since it cannot be done, women can set the time of gas extraction and defecation as time/date; they'll record it. Assessment of pain level, first 8. After the time of 16 and 24. in the hours will be made.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: chewing gum Group — control of consciousness chewing gum listening to bowel sounds assessment of pain
  Arms: chewing gum Group
Procedure: Control group — control of consciousness listening to bowel sounds assessment of pain
  Arms: Control group

SUMMARY:
Surgical interventions, such as restoring the health of patients and eliminating their existing symptoms, the surgical process can have many negative effects on the patient. In order to minimize these complications, the Accelerated Recovery Protocol After Surgery (ERAS) has also found widespread use in obstetric surgery. The ERAS protocol consists of different evidence-based practices at each stage, before, during, and after surgery. Stool and gas extraction, especially colorectal reported that chewing gum has a positive impact on the time/ can be used after pelvic surgical procedures, perioperative care guide contains reported in ERAS protocols, evidence-based, inexpensive, easily applied, and easily tolerated a practice that is emphasized.

DETAILED DESCRIPTION:
Surgical interventions, such as restoring the health of patients and eliminating their existing symptoms, the surgical process can have many negative effects on the patient. In order to minimize these complications, the Accelerated Recovery Protocol After Surgery (ERAS) has also found widespread use in obstetric surgery. The ERAS protocol consists of different evidence-based practices at each stage, before, during, and after surgery. Stool and gas extraction, especially colorectal reported that chewing gum has a positive impact on the time/ can be used after pelvic surgical procedures, perioperative care guide contains reported in ERAS protocols, evidence-based, inexpensive, easily applied, and easily tolerated a practice that is emphasized. Different studies have been conducted to determine the effect of chewing gum on intestinal peristalsis. Intestinal sounds and defecation of chewing gum after cesarean section surgery. A limited number of studies on patients with total laparoscopic hysterectomy exist on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Total laparoscopic hysterectomy is the most common type of hysterectomy.,

  * Who is literate,
  * over 18 years old,
  * The body mass index is dec 18.50-24.99 kg/m2,
  * Able to communicate, no language problems.
  * No history of allergies,
  * Who volunteered to participate in the study and received my approval,
  * No complications during the operation,
  * With a patient who is not diagnosed with a mental and psychiatric illness

Exclusion Criteria:

* Who can not adapt to the treatment process,

  * Developing postoperative complications,
  * Chemotherapy - receiving radiation therapy therapy,
  * With epilepsy disease,
  * With any history of allergies,
  * A history of dental and gum diseases, with difficulty chewing,
  * With a problem of the mucous membrane inside the mouth,
  * Using drugs that can affect bowel function due to systemic diseases,
  * Patients with a mental disability or a perception problem

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change of the postoperative baseline bowel activity (bowel sounds) at the first 6 hours postoperative pain after total laparoscopic hysterectomy | within postoperative first 6 hours, three times per 2 hours
  Time to first detection of postoperative bowel activity will be evaluated by the same healthcare worker via physical examination (oscultation of the four quadrants)

CONTACTS AND LOCATIONS:
Overall Officials: Melike Dissiz, Professor, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT05135416/ICF_000.pdf